CLINICAL TRIAL: NCT05031832
Title: The Interrelationship Between Chemsex Engagement and HIV Biomedical Prevention in MSM
Brief Title: Chemsex Engagement and HIV Biomedical Prevention in MSM
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ngai Sze WONG, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: MSS344R
Record Dates: First submitted 2021-08-30; First posted 2021-09-02 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Recreational Drug Use
Keywords: Chemsex engagement; Pre-exposure prophylaxis; Antiretroviral therapy; men who have sex with men
MeSH Terms: conditions — Recreational Drug Use; Homosexuality | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV-negative
  Interventions: Diagnostic Test: HIV test
- HIV-positive

INTERVENTIONS:
Diagnostic Test: HIV test — HIV test would be offered to self-reported HIV-negative / unknown HIV status MSM to confirm their HIV status
  Groups: HIV-negative

SUMMARY:
HIV biomedical prevention through treatment-as-prevention (TasP) and pre-exposure prophylaxis (PrEP) is highly efficacious for reducing HIV transmission risk. The benefits could be undermined by the rising HIV transmission risks in men who have sex with men (MSM) who engaged in chemsex. This project aims to assess the impacts of chemsex on the growth of the HIV epidemic by exploring the complex relationships between chemsex engagement and usage of HIV biomedical prevention in MSM in Hong Kong. Participants would be recruited from the community and clinics in 2 cross-sectional studies (500 HIV-negative and 500 HIV-positive MSM), for HIV self-testing and completing an electronic questionnaire. The association of chemsex would be examined between PrEP-naïve and PrEP experienced HIV-negative MSM, and between good and poor adherence to antiretroviral therapy (ART) among HIV-positive subjects in case-control analyses using logistic regression and multilevel models. The main outcomes include coverage of biomedical prevention in MSM, and their drug use patterns.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* male
* have had sex with men since 2019
* could be communicated in English or Chinese

Exclusion Criteria:

* failed to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sexually active adult men who have sex with men living in Hong Kong, and able to complete the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
pre-exposure prophylaxis coverage | 6 months
  proportion of HIV-negative MSM taking pre-exposure prophylaxis; based on self-reported data in questionnaire
Good antiretroviral therapy adherence | 2 years
  proportion of HIV-positive MSM with good antiretroviral therapy adherence; based on self-reported data (CD4 count, viral load level, history of stoppoing ART / missing doses) in questionnaire
Drug use pattern | 6 months
  types of drugs taken for chemsex engagement (taking before or during sex); based on self-reported data in questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No